CLINICAL TRIAL: NCT06869863
Title: Open Single-center Study of Tolerability, Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of the Medicinal Product MediReg® (Human Mesenchymal Stromal Cell Secretome), Lyophilizate for Preparation of Solution for Injection in Patients with Severe Spermatogenesis Disorders
Brief Title: Study of Tolerability, Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of the Medicinal Product MediReg®
Acronym: MARS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lomonosov Moscow State University Medical Research and Educational Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSU 001
Record Dates: First submitted 2025-02-10; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Azoospermia, Nonobstructive; Teratospermia; Oligospermia; Men Infertility
Keywords: men infertility; azoospermia
MeSH Terms: conditions — Azoospermia, Nonobstructive; Teratozoospermia; Oligospermia; Azoospermia | interventions — Injections; Clomiphene

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, open-label, uncontrolled phase I/II study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of the medicinal product MediReg® (Human Mesenchymal Stromal Cell Secretome), lyophilizate for preparation of solution for injection will be performed in patients with severe forms of spermatogenesis disorders manifested as severe oligoasthenoteratozoospermia (OAT), non-obstructive azoospermia, high sperm DNA fragmentation (30% and more).
  The absence of a comparison group is due to the fact that participation in the study carries a risk to patients that exceeds the minimum risk, Out of 60 patients, 20 subjects will be treated with MediReg® with evaluation of pharmacokinetics before and after drug administration.
  To confirm the non-randomization of the recorded changes, a control group receives therapy according to the approved recommendations, spermogram and hormonal profile assessment on days 0...90 is provided
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MediReg (Experimental): 60 patients (20 patients in first phase of the study and 60 patients in 2nd phase) a single injection of 0.5 ml of the investigational drug intratesticularly under the white membrane, alternately in both testicles
  Interventions: Biological: Medicinal product MediReg® (Human Mesenchymal Stromal Cell Secretome), lyophilizate for preparation of solution for injection in patients with severe spermatogenesis disorders
- Clomiphene /Triovit,/Folic acid (Active Comparator): Clostilbegit (clomiphene) 50 mg 1 tablet x 1 p a day - 3 months, Triovit - 1 tablet x 1 p a day - 3 months, Folic acid - 1 tablet x 1 p a day - 3 months.
  Interventions: Other: Clostilbegit (clomiphene) 50 mg 1 tablet x 1 p a day - 3 months, Triovit - 1 tablet x 1 p a day - 3 months, Folic acid - 1 tablet x 1 p a day - 3 months.

INTERVENTIONS:
Biological: Medicinal product MediReg® (Human Mesenchymal Stromal Cell Secretome), lyophilizate for preparation of solution for injection in patients with severe spermatogenesis disorders — Human mesenchymal stromal cell secretion1 containing vascular endothelial growth factor (VEGF)2 ≥ 5,0 нг
  Arms: MediReg
Other: Clostilbegit (clomiphene) 50 mg 1 tablet x 1 p a day - 3 months, Triovit - 1 tablet x 1 p a day - 3 months, Folic acid - 1 tablet x 1 p a day - 3 months. — Combination treatment recommended by standards
  Arms: Clomiphene /Triovit,/Folic acid

SUMMARY:
The study is open to patients with severe forms of male infertility (non-obstructive disorders of spermatogenesis, including azoospermia).

The Phase I/II clinical trial is being conducted at the Lomonosov Moscow State University and is aimed at studying the efficacy and safety of the innovative drug "MediReg® (Human Mesenchymal Stromal Cell Secretome)", lyophilizate for preparation of solution for injection, 1.0 ml/dose for treatment of male infertility. The study was approved by the Ministry of Health of the Russian Federation. The study is planned to include men aged 21 to 60 years with severe spermatogenesis disorders manifested as severe oligoasthenoteratozoospermia (OAT), non-obstructive azoospermia, high sperm DNA fragmentation (30% and more) and faced with the inability to conceive, including with the help of assisted reproductive technologies within 12 months from the date of diagnosis The aim of the therapy is to improve the spermogram indicators in order to increase the chances of successful use of assisted reproductive technologies.

The drug is injected once under the protein sheath of both testicles. Observation in 1 week after the drug administration is carried out in hospital. Follow-up is performed by outpatient visits to the research center.

The clinical trial is planned to enroll at least 80 adult patients aged 21 to 60 years with severe spermatogenesis disorders The study will include 3 periods:Screening Period - Day -15...0.

, Period of study drug administration and inpatient follow-up - Day 1 through Day 7., Follow-up period - through Day 90.

The total duration of participation in the study, including the screening period and the follow-up period, will not exceed 119 days. After the end of the study period, the study will be followed up for 1 year to record delayed adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male patients aged 21-60 years at the time of inclusion in the study. 2. Persistent severe disorders of spermatogenesis, manifested as severe oligoasthenoteratozoospermia (OAT)*, non-obstructive azoospermia, high sperm DNA fragmentation (30% or more), including those caused by secretory infertility according to dynamic control of spermogram (at least 12 months from the moment of inclusion in the study).

  * "Persistent severe OAT" should be considered as disorders when sperm concentration <5 million/mL, progressively motile sperm <13% and/or total number of progressively motile sperm in the ejaculate (PMPM) <5 million, with the proportion of normal sperm <1% according to the dynamic control of spermogram (at least 12 months from the moment of inclusion in the study).

    3. inability to conceive against the background of "severe forms" of male infertility, not amenable to treatment, including assisted reproductive technologies, within 12 months from the moment of diagnosis or refusal to use assisted reproductive technologies.

    4. Voluntarily signed Informed consent by the patient to participate in the clinical trial.

    5. Willingness of patients and their sexual partners to use reliable contraceptive methods (combination of at least 2 methods, including 1 barrier method, e.g., use of spermicide and condom) from the time of signing the informed consent until at least 1 month after completion of study participation.

    6. Patient willingness to follow all the requirements of the Protocol.

Exclusion Criteria:

* 1. Age younger than 21 and older than 60 years at the time of inclusion in the study.

  2. developmental anomalies of the genitourinary system (according to bladder and kidney ultrasound).

  3. surgical interventions on genitourinary organs in the history, except for surgical interventions associated with assisted reproductive technologies. 4.

  4. Systemic diseases requiring administration of corticosteroids, cytostatics, radiation therapy.

  5. Inflammatory diseases of the urinary and/or reproductive system. 6. Infectious diseases (including STDs) of the urinary and/or reproductive system.

  7. Hereditary factors of infertility: (Klinefelter syndrome (all variants), autosomal abnormalities (all variants), carrying the cystic fibrosis gene (all variants), presence of Y-chromosome microdeletions (all AZF variants), autosomal defects with severe phenotypic abnormalities and infertility (Prader-Willi, Bardet-Biedl, Noonan syndromes, myotonic dystrophy, dominant polycystic kidney disease, 5-alpha-reductase enzyme deficiency, etc.). д.).

  8. Obstructive azoospermia by history or established by screening examination. 9. Positive test for HIV, hepatitis B and C, syphilis. 10. Severe liver failure or active liver disease (transaminase activity exceeding 5 times the upper limit of the local laboratory norm).

  11. Renal dysfunction with serum creatinine levels exceeding 120 µmol/L. 12. Cardiovascular diseases in the history within 6 months before inclusion in the study, such as myocardial infarction, angina pectoris, severe ventricular arrhythmia, heart failure (NYHA class II-IV).

  13. Neurologic (Parkinson's disease) and/or psychiatric illnesses with a history or established by screening examination.

  14. Cancer with a history of cancer or as determined by screening examination (as determined by OBP and renal ultrasound, bladder ultrasound, prostate TRUS).

  15. Hypersensitivity to any of the components of the study drug in the history. 16. Mental illness, severe cognitive impairment, need to take tranquilizers, neuroleptics and/or antidepressants during this study.

  17. Severe somatic illnesses that, in the opinion of the investigator, may affect the patient's safety and ability to comply with the Protocol.

  18. A history of drug dependence. 19. Positive urinalysis for psychotropic and narcotic drugs, psychoactive medications.

  20. Intake of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to 1⁄2 liter of beer, 200 ml of wine, or 50 ml of alcohol) or a history of alcoholism.

  21. Detection of alcohol vapor in breath 22. Participation in another clinical trial currently or in the previous 30 days prior to the screening visit.

  23. Patient's inability to understand or comply with study procedures or patient's refusal to cooperate with a particular investigator

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Semen Analysis | 90 days
  In more than 30% of patients with nonobstructive azoospermia appearance of sperm cells in semen

SECONDARY OUTCOMES:
Increase in inhibin B level by more than 20% from baseline | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Okhobotov, doctor of sciences, Principal Investigator — University Clinic of the Medical Scientific and Educational Institute of Moscow State University named after M.V.Lomonosov, Moscow,; Anastasia Efimenko, doctor of sciences, Study Chair — University Clinic of the Medical Scientific and Educational Institute of Moscow State University named after M.V.Lomonosov, Moscow, Moscow 119234
Locations (1):
- University Clinic of the Medical Scientific and Educational Institute of Moscow State University named after M.V.Lomonosov, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No